CLINICAL TRIAL: NCT04352309
Title: REAl World Evidence Of The Effectiveness And Clinical Practice Use Of Glecaprevir/Pibrentasvir For 8 Weeks Treatment In Patients With Chronic HepatitiS C GenotYpes 1 to 6 And Liver Cirrhosis In Russian Federation (EASY)
Brief Title: Efficacy Study Of Oral Glecaprevir/Pibrentasvir Tablet In Pediatric (12 Years and Older) And Adult Treatment-Naive Participants With Chronic Hepatitis C Genotypes 1 To 6 And Liver Cirrhosis
Acronym: EASY
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-276
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: HCV, Hepatitis C Virus; Hepatitis C; Liver Cirrhosis; GLE/PIB
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Treated With Glecaprevir/Pibrentasvir (GLE/PIB): Participants will receive GLE/PIB over 8 weeks of therapy as prescribed by their physicians.

SUMMARY:
Hepatitis C Virus (HCV) infection is among the most common of all chronic liver diseases. HCV predominantly affects liver cells and causes the liver to become inflamed and damaged. This can lead to cirrhosis (scarring of the liver) and liver cancer leaving trial participants with need for liver transplant. The purpose of this study is to see how effective Glecaprevir/Pibrentasvir (GLE/PIB) is in a real world setting of participants with chronic HCV genotypes 1 to 6 and liver cirrhosis who have never received any treatment for HCV.

GLE/PIB is a drug developed for the treatment of HCV infection. This is a prospective (future), observational study in treatment-naive (those who have not received treatment) participants with HCV genotypes 1 to 6 and compensated cirrhosis. All study participants will receive GLE/PIB as prescribed by their study doctor in accordance with approved local label. Pediatric (12 years and older) and adult participants with a diagnosis of HCV genotypes 1 to 6 and compensated cirrhosis will be enrolled in the study in Russian Federation.

Participants will receive GLE/PIB tablets to be taken by mouth daily according to their physicians' prescription. The total duration of the study is 20 weeks, with a treatment period of 8 weeks and a follow up period of 12 weeks.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice and participants will be followed for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve male or female with confirmed CHC, genotypes 1, 2, 3, 4, 5, or 6, with compensated liver cirrhosis, receiving combination therapy with the all oral GLE/PIB regimen for 8 weeks according to standard of care, international guidelines and in line with the current local label.
* Participants may be enrolled up to 4 weeks after treatment initiation.

Exclusion Criteria:

* Participating or intending to participate in a concurrent interventional therapeutic trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Treatment-naive Pediatric (12 years and older) and adult participants with confirmed Chronic Hepatitis C (CHC), genotypes 1, 2, 3, 4, 5, or 6 with compensated cirrhosis, being treated with oral Glecaprevir/Pibrentasvir (GLE/PIB) according to standard of care, international guidelines and in line with the current local label.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Percentage Of Participants Achieving Sustained Virologic Response At 12 Weeks (SVR12) | At Week 20
  SVR12 is defined as Hepatitis C Virus (HCV) RNA < 50 IU/ml or < lower limit of quantification/detection (LLoQ/D) available at the site 12 weeks (i.e.,>=70 days) after the last actual dose.

SECONDARY OUTCOMES:
Number Of Participants Achieving SVR12 After Last Actual Dose Of GLE/PIB At 12 Weeks In Subgroups Of Interest | At Week 20
  SVR12 is defined as HCV RNA < lower limit of quantification/detection (LLoQ/D) 12 weeks (i.e., >=70 days) after the last actual dose of GLE/PIB with a sensitive polymerase chain reaction (PCR) available in the clinical site in the settings of the Russian Federation in subgroups of interest.
Number Of Participants With Co-morbidities | At Week 20
  Participants who have other existing medical conditions.
Number Of Participants Taking Concomitant Medication | At Week 20
  Participants who take other medications along with Glecaprevir/Pibrentasvir (GLE/PIB).
Percentage Of GLE/PIB Dose Taken In Relation To The Prescribed Target Dose | At Week 20
  Percentage of GLE/PIB dose taken by participant report in relation to the prescribed target dose (number of pills taken out of the number that should have been taken).
Number of Participants With Adverse Events | Baseline (Week 0) To 30 days post last dose
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug. A Serious Adverse Event ( SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Percentage of Participants With Shifts in Clinical Laboratory Values | Baseline (Week 0) to Week 20
  Percentage of participants with clinically significant change in laboratory parameters of interest (hematology, biochemistry, virology, coagulation, and urinalysis), post-baseline during treatment, will be summarized.
Number Of Health Care Resource Utilization (HCRU) Over Time Overall And By Subpopulations Of Interest | At Week 20
  HCRU for a participant will be the total number of visits/touchpoints (face to face or phone call) with a Health Care Professional (HCP) or designee in relation to their Hepatitic C Virus (HCV) infection during the study.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (6):
- Russia (6):
  - South Ural State Medical University /ID# 225501, Chelyabinsk
  - Irkutsk Regional Center for the Prevention and Control of AIDS and Infections /ID# 225499, Irkutsk
  - S. P. Botkin City Hospital /ID# 225500, Oryol
  - Samara Region Clinical HIV/AIDS Prevention and Control Center /ID# 222582, Samara
  - Stavropol State Medical University /ID# 226589, Stavropol
  - Medical center Academy /ID# 226587, Ulyanovsk

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P20-276&Latitude=&Longitude=&LocationName=#additional-resources-section